CLINICAL TRIAL: NCT07191782
Title: Examining the Efficacy of the PRAISE With Coaching Program in Reducing Peer Aggression and Bullying
Brief Title: Examining the Efficacy of the PRAISE With Coaching Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: The School District of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-022385; 1R49CE003566-01-00 (Other Grant/Funding Number: CDC); 1R49CE003566-01 (NIH)
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Aggression Childhood; Bullying Victimization; Social Behavior
Keywords: late elementary school; universal classroom-based; aggression prevention; bullying prevention; relational aggression; coaching
MeSH Terms: conditions — Social Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison Schools (No Intervention): These schools do not receive the PRAISE intervention. These schools can have their standard aggression and bullying practices such as community meeting, restorative circles, Second Step program, and the Olweus program. We will measure what classrooms in the comparison condition are doing, but we will not intervene.
- Intervention Schools (Experimental): These schools will receive the PRAISE program which includes training and coaching from the research team.
  Interventions: Behavioral: Universal, classroom-based, Bullying and Aggression Prevention Program

INTERVENTIONS:
Behavioral: Universal, classroom-based, Bullying and Aggression Prevention Program — PRAISE is a universal, classroom-based aggression and bullying prevention program that addresses all forms (physical, verbal, relational, cyber), with a strong focus on the relational and reactive behaviors. All emotional and social skills taught focus on applying and practicing the skills within peer relationships. This program has gone through iterative development and adaptations using a community-based participatory approach whereby the elementary students and staff were active partners with researchers in refining the program. Specific attention was paid to ensuring that the program is feasible for schools to implement and sustain while also being relevant and relatable for students from a variety of backgrounds and school communities (e.g., under-resourced, higher levels of community violence). This updated PRAISE includes ~14 sessions (amounts can vary by grade) and training and coaching for school-based facilitators of the program.
  Arms: Intervention Schools

SUMMARY:
The PReventing Aggression In Schools Everyday (PRAISE) Program has evidence of impact when run by research staff. PRAISE was adapted using community-based participatory research to a coaching model whereby school-staff are trained to facilitate the program and receive ongoing coaching from research staff. The overall objective is to demonstrate the efficacy of the adapted PRAISE program when facilitated by in-school staff.

DETAILED DESCRIPTION:
PRAISE is an aggression and bullying prevention program that includes curriculum to help 3rd through 5th graders learn skills to identify feelings, use calming-down strategies, interpret others' intentions accurately, and consider choices when responding to conflict. PRAISE also has lessons on increasing empathy and perspective-taking, and empowering students to be positive bystanders.

Using a randomized control trial of at least 8 elementary schools (3rd-5th grade) we will examine 2 aims:

Aim 1: Examine the efficacy of PRAISE at reducing students' peer aggression and bullying and improving social problem-solving skills, positive bystander behaviors, and self-efficacy for non-violence.

Aim 2. Examine the moderating role of implementation and student- and facilitator-related factors on the main outcomes of interest.

ELIGIBILITY:
Student Inclusion Criteria:

* Enrolled in one of the participating school sites
* In a 3rd-5th grade classroom participating in the study

Staff Inclusion Criteria:

* Employed by one of the participating school sites
* Teach and/or provide services to students in 3rd-5th grade

Students Exclusion Criteria:

* Do not speak English
* Special education students not integrated in a regular education classroom
* Student not in Grades 3-5 at the participating school sites

Teacher Exclusion Criteria:

* Do not speak English
* Do not teach/provide services with 3rd-5th grade students at the participating school sites

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1008 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Peer Ratings of Peer Aggression | At baseline and post intervention, approximately 8 months.
  Measured via peer-reports. Students rate the frequency that each classmate engages in relational (1 item), verbal (1 item) and physical (1 item) aggression on a scale from 1- Not at All to 5- A Whole Lot. Each individual child gets an average score based the classroom peer reports with higher scores reflecting more of that outcome.
Knowledge of Social Information Processing | At baseline and post intervention, approximately 8 months.
  Student self-report of social information processing knowledge will be gathered using the Knowledge of Anger Problem Solving measure (9 items) where items are scored a 1 if correct and 0 if incorrect and summed (Range: 0-9), higher scores reflect better social information processing
Hostile Attributions | At baseline and post intervention, approximately 8 months.
  Student self-report of hostile attributions will be assessed using the Cartoon-Based Hostile Attributional Bias measure, with 2 relational vignettes and 2 physical vignettes, with one question asking whether a behavior was intentional or unintentional. Each vignette has a range of 0 (no bias) to 4 (strong bias). Scores on the 2 items per vignette type (relational, physical) are summed where higher scores reflect a worse outcome.
Self-efficacy for Non-Violence | At baseline and post intervention, approximately 8 months.
  Student self-report of their use of non-aggressive or violent responses when in a conflict with a peer will be assessed using 9 items drawn from the measure developed for the Multisite Violence Prevention Project with a range of 1-Not at to 4-Very confident. Items are averaged with higher scores reflecting more conference in their ability to not use violent or aggressive responses.
Reactive/proactive Aggression | At baseline and post intervention, approximately 8 months.
  Measured via student self-report using items drawn from the Peer Conflict Scale -Youth Version measure, the proactive relational (6 items) and reactive relational (6 items) and overt (5 items). Items, with a range of 1-Not at all true to 4-Definitely true, will be averaged per scale. Higher scores indicate more proactive relational, reactive relational and reactive overt aggression.
Bullying Perpetration | At baseline and post intervention, approximately 8 months.
  Bullying will be assessed using the Behavior Based Bullying measure (9 items; Range: 1- Never to 4- or more times per month), items are averaged where higher scores means more bullying perpetration.
Cyberbullying | At baseline and post intervention, approximately 8 months.
  Student Self-report on items drawn from the European Cyberbullying Intervention Project Questionnaire will assess two scales: cyberbullying perpetration (7 items) and victimization (7 items) with answers ranging from 1-Never to 5-A few times a week. Items will be averaged such that higher score is more perpetration or victimization experiences.
Bystander Behaviors | At baseline and post intervention, approximately 8 months.
  Self-report of positive bystander behaviors will be assessed using 5 items drawn from the Maryland Safe and Supportive Schools (MDS3) Climate Survey with answers ranging from 1-Never to 5-All the time. Items are averaged with higher scores indicating more use of positive bystander behaviors.
Relational and Overt Aggression | At baseline and post intervention, approximately 8 months.
  Using teacher report on each child in their classroom, the Children's Social Behavior Questionnaire will assess a child's relational (7 items) and overt (4 items) aggression with a range of 1-Never true to 5-Almost always true. Items are averaged per scale with higher scores indicating more relational or overt aggression.

SECONDARY OUTCOMES:
Empathy | At baseline and post intervention, approximately 8 months.
  Student self-report of cognitive empathy using the perspective taking scale of the Interpersonal Reactivity Index (6 items; Range: 1-Never to 5-All the Time). Items are averaged where higher scores indicated more empathy.
Peer Bullying-Victimization | At baseline and post intervention, approximately 8 months.
  Student self-report of victimization by peers using the Social Experience Questionnaire (SEQ; 10 items, Range: 1-Never to 5-All the time). Items are averaged with higher scores indicated more peer bullying-victimization experiences.
Academic Engagement | At baseline and post intervention, approximately 8 months.
  Teacher report on each child in their classroom will be used to assess academic engagement using the Academic Competence Evaluation Scale (8 items; Range: 1-Never to 5-Almost Always). Items are averaged with higher scores reflecting more engagement.
Student-teacher Relationship | At baseline and post intervention, approximately 8 months.
  Teacher report on each child in their classroom of their perceived relationships (closeness and conflict) using the Closeness (5 items) and Conflict (5 items) drawn from the Student Teacher Relationship Scales (STRS; Range: 1-Definitely doesn't apply to 5-Definitely applies). Items per scale are averaged such that higher scores indicated more closeness or conflict between teacher and student.
Class Climate | At baseline and post intervention, approximately 8 months.
  Student self-report of their perception of the class academic and social climate using 6 items drawn from the Maryland Safe and Supportive Schools (MDS3) Climate Survey with a range from 1-Strongly Agree to 4-Strongly Disagree. Items are averaged such that higher scores indicate a more positive classroom climate.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy E Waasdorp, PhD MSEd, Principal Investigator — Children's Hospital of Philadelphia; Brooke S Paskewich, Psy.D, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No